CLINICAL TRIAL: NCT00678353
Title: Prospective Data Collection From the Stryker Biotech Pivotal IDE Study of OP-1 Putty in Uninstrumented Posterolateral Fusions
Brief Title: Study of OP-1 Putty in Uninstrumented Posterolateral Fusions
Status: Completed | Type: Observational
Sponsor: Olympus Biotech Corporation (Industry)
Responsible Party: Shinichi Torii, Olympus Biotech
Other Study IDs: 06-UPLF-01
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Degenerative Lumbar Spondylolisthesis
Keywords: Degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Follow-up to S01-01US, conducted to expand information

SUMMARY:
This study is to provide additional data to support the safety and efficacy of OP-1 Putty as a replacement for autograft in patients undergoing posterolateral spinal fusion.

DETAILED DESCRIPTION:
Follow-up study 06-UPLF-01 was a prospective collection of longer-term data on the patient population from pivotal study S01-01US, and was conducted to expand the information regarding efficacy, particularly with regard to radiographic assessment of fusion, as well as the longer-term safety of OP-1 Putty in uninstrumented posterolateral fusion (PLF) as compared to autograft

ELIGIBILITY:
Inclusion Criteria:

1. The patient was treated in Stryker Biotech clinical protocol S01-01US (Pivotal IDE study) and not a retreatment failure at the time of completion.
2. The patient or legal guardian is willing and able to understand, sign and date the study specific Patient Informed Consent.
3. The patient agrees to complete the necessary clinical and radiographic evaluations.

Exclusion Criteria:

1. There are no exclusion criteria for participation in this protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in clinical protocol S01-01US
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Evidence of bone by CT scan | 3+ years post-treatment from the Pivotal study S01-01US

SECONDARY OUTCOMES:
Re-assessments of all clinical parameters from S01-01US | 3+ years post-treatment from the Pivotal study S01-01US

CONTACTS AND LOCATIONS:
Locations (22):
- United States (19):
  - Santa Monica, California
  - Stanford, California
  - Denver, Colorado
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Chicago, Illinois
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Akron, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Fairfax, Virginia
- Canada (3):
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario